CLINICAL TRIAL: NCT03007043
Title: Genetic Variation in Gonadotropin and Gonadotropin Receptor Genes as a Causative Factor of Suboptimal Response Following Ovarian Stimulation for IVF/ICSI. A Prospective Cohort Study
Brief Title: Genetic Variation in Gonadotropin and Gonadotropin Receptor Genes and Suboptimal Response
Status: Completed | Type: Observational
Sponsor: Fundacion Dexeus (Other)
Responsible Party: Principal Investigator, Nikolaos Polyzos, Professor, Fundacion Dexeus
Other Study IDs: 2016.Polymorphisms_COS
Record Dates: First submitted 2016-12-28; First posted 2016-12-30 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Fertility Disorders
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal responders: Normal response following IVF
  Interventions: Other: blood sample
- Suboptimal responders: Suboptimal response following IVF
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample

SUMMARY:
To evaluate the difference in the prevalence of the main FSHR polymorphism (ASN680Ser), as well as other, less studied, gonadotropin polymorphisms between ovarian response groups, following ovarian stimulation

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-38 years old
2. BMI 18-28
3. Antral follicle count (AFC) > 9 or Anti-mullerian hormone (AMH) >1.1 ng/ml
4. 1st or 2nd ovarian stimulation cycle for IVF/ICSI
5. Planned to undergo ovarian stimulation with 150IU of rFSH in a fixed GnRH antagonist protocol

Exclusion Criteria:

1. Antral follicle count (AFC) <9 and AMH<1.1 ng/ml
2. PCOS patients according to the Rotterdam criteria
3. Patients undergoing in vitro maturation (IVM)
4. Untreated endocrine abnormalities

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile women undergoing ovarian stimulation
Sampling Method: Probability Sample
Enrollment: 364 (Actual)
Dates: Start 2016-11; Primary Completion 2019-04 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
prevalence of the main FSH receptor polymorphism | 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- Dexeus Salud de la Mujer, Barcelona, Spain
- Department of Obstetrics and Gynecology, University of Medicine and Pharmacy HCMC, Ho Chi Minh City, Vietnam and Research Center for Genetics and Reproductive Health (CGRH), School of Medicine, Vietnam National University HCMC, Ho Chi Minh City, Vietnam

REFERENCES:
- [Derived] Neves AR, Vuong NL, Blockeel C, Garcia S, Alviggi C, Spits C, Ma PQM, Ho MT, Tournaye H, Polyzos NP. The effect of polymorphisms in FSHR gene on late follicular phase progesterone and estradiol serum levels in predicted normoresponders. Hum Reprod. 2022 Oct 31;37(11):2646-2654. doi: 10.1093/humrep/deac193. PMID 36069495
- [Derived] Polyzos NP, Neves AR, Drakopoulos P, Spits C, Alvaro Mercadal B, Garcia S, Ma PQM, Le LH, Ho MT, Mertens J, Stoop D, Tournaye H, Vuong NL. The effect of polymorphisms in FSHR and FSHB genes on ovarian response: a prospective multicenter multinational study in Europe and Asia. Hum Reprod. 2021 May 17;36(6):1711-1721. doi: 10.1093/humrep/deab068. PMID 33889959